CLINICAL TRIAL: NCT05619822
Title: A Comprehensive Third-generation Intervention for People With Psychosis and Post-traumatic Stress Symptoms; Design, Implementation and Effectiveness
Brief Title: A Comprehensive Third-generation Intervention for People With Psychosis and Post-traumatic Stress Symptoms
Acronym: IITG-PPT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCHIZO
Record Dates: First submitted 2022-10-26; First posted 2022-11-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Trauma, Psychological; Psychosis
Keywords: Psychosis; Trauma; Psychological Intervention; EMDR
MeSH Terms: conditions — Psychological Trauma; Psychotic Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + waiting list (Other): Treatment as usual
  Interventions: Behavioral: TAU
- TAU + A comprehensive third-generation intervention (Experimental): he protocol will bedeveloped following the three stages of recovery from trauma (Herman, 2015): first, focusing on establishing the therapeutic alliance and safety; second, focusing on recounting and re-processing the traumatic event; and third, focusing on reconnecting with others and with life despite the trauma experienced. The therapy will be administered in 11 90-minute individual sessions per week, combining strategically ACT, Mindfulness, EMDR as well as Positive Psychology interventions.
  Interventions: Behavioral: TAU + A comprehensive third-generation intervention

INTERVENTIONS:
Behavioral: TAU + A comprehensive third-generation intervention — This is a individual intervention with with a total of 12 sessions: Session 1. Constructing the Therapy Experience. Session 2. Life history and immediate reactions to trauma. Session 3. Preparing to deal with trauma. Session 4. Regulating emotions. Session 5-9. Focusing on retelling and processing the traumatic event (EMDR PHASES_PHASE 3: Evaluation of the traumatic memory. EMDR PHASE 4: Desensitization. EMDR PHASE 5: Positive Belief Installation. PHASE 6: Body Scan). Session 9. Re-evaluating traumatic memory and self-care through positive emotions. Session 10. Cultivating self-kindness. Session 11. Developing a healthy identity. Session 12. Building a better future
  Arms: TAU + A comprehensive third-generation intervention
Behavioral: TAU — Treatment as usual
  Arms: TAU + waiting list

SUMMARY:
Existing data suggest that both trauma and Post-Traumatic Stress Disorder (PTSD) are very common among individuals with psychosis. The presence of PTSD symptoms in psychosis is associated with worse clinical outcomes and poorer social functioning. However, PTSD is a poorly attended and poorly studied condition among this population. Research to date indicates that trauma-focused treatments are safe and effective for PTSD, even when psychotic comorbidity is present. Recent systematic reviews of psychological interventions for trauma in psychosis found that are effective in reducing trauma symptoms, suggesting that they should be implemented in front-line services. Nonetheless, larger confirmative trials are required to form robust conclusions.The aim of this project is to examine the efficacy of comprehensive third-generation protocol for people with comorbid trauma and psychosis.

DETAILED DESCRIPTION:
This study is a randomized clinical trial at psychiatric rehabilitation services of the Public Network of Care for people with serious mental disorders. We hypothesize that participants receiving the intervention, in comparison with controls, will show a reduction in general, PTSD and psychotic symptomatology, an improvement in levels of functioning and well-being, a greater ability to regulate emotions with more help-seeking behaviours.

Given the complexity of both psychosis and PTSD and the reluctance of professionals to treat it, we plan to develop a precise comprehensive protocol. In order to address all issues associated with both psychosis and comorbid PTSD, the protocol will be developed following the three stages of recovery from trauma: first, focusing on establishing the therapeutic alliance and safety; second, focusing on recounting and re-processing the traumatic event; and third, focusing on reconnecting with others and with life despite the trauma experienced. The therapy will be adapted to the characteristics of people with SMD and administered in 11 90-minute individual sessions per week, combining strategically ACT, Mindfulness, EMDR as well as Positive Psychology interventions.

ELIGIBILITY:
Inclusion Criteria:

Those showing a high risk of PTSD (TSQ ≥6) will be further evaluated to determine whether they meet the inclusion criteria. Participants must:

* Be between the ages of 18 and 65 fluent enough in Spanish language;
* Meet the criteria for a diagnosis of a psychotic spectrum disorder or a mood disorder with psychotic symptoms according to MINI (Sheeman et al., 1997);
* Meet PTSD diagnostic criteria according to the Clinician-Administered PTSD Scale (CAPS; Blake et al., 1995)

Exclusion Criteria:

* Those who have a diagnosis of substance or alcohol abuse or dependence in the 30 days prior to participation in the study
* To have a severe neurocognitive problems or brain damage that interfere with the basic processing of information in psychotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from posttraumatic symptoms at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  International Trauma Questionnaire (ITQ; Cloitre, et al., 2018).Higher scores mean a worse outcome.
Change from psychotic symptoms at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  Psychotic Symtoms Rating Scale (Haddock et al., 1999).Higher scores mean a worse outcome.
Change from psychopathological symptoms at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  Symptom Checklist 45-SCL-90_r brief (Davison et al., 1997). Higher scores mean a worse outcome.
Change from dissociative symptoms at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  The Dissociative Experience Scale Taxon (DES-T; Waller & Ross, 1997). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from Personal and Social functioning at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  Personal and Social Performance Scale (PSP; Morosini y cols., 2000). Higher scores mean a worse outcome.
Change from Wellbeing at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  Scales of Psychological Well-Being (SPWB; Ryff & Keyes,1995). Higher scores mean a better outcome.
Change from satisfaction with life at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  Satisfaction with Life Scale (SWLS; Diener et al., 1985). Higher scores mean a better outcome.
Change from Attachment at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  Psychosis Attachment Measure (PAM; Berry et al., 2006; Sheinbaum et al., 2013). Higher scores mean a worse outcome.
Change from Emotion Regulation at 12 weeks and 6 months | Change baseline, 12 weeks, and 6 months
  Cognitive Emotion Regulation Questionnaire (CERQ; Garnefski & Kraaij, 2007). Higher scores mean a worse outcome for disfunctional dimensions and a better outcome for functional dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Valiente, Ph.D., Principal Investigator — Universidad Complutense de Madrid; Regina Espinosa, Ph.D., Principal Investigator — Universidad Camilo Jose Cela
Locations (1):
- Carmen Valiente, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code